CLINICAL TRIAL: NCT03299153
Title: The Effects of Barberry Juice Consumption on Glycaemic Control, Lipid Profile, Blood Pressure and Oxidative Stress in Patients With Type 2 Diabetes: A Randomized Clinical Trial
Brief Title: The Effects of Barberry Juice Consumption in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, National Nutrition and Food Technology Research Institute, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1534
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients in this group were received 200 ml/d barberry juice for tow month
  Interventions: Other: barberry juice
- control group (No Intervention): patients in this group received no intervention

INTERVENTIONS:
Other: barberry juice
  Arms: Intervention group

SUMMARY:
The aim of this study was to investigate the effect of barberry juice (BJ) as a natural antioxidant, on cardiovascular risk factors in patients with type 2 diabetes (T2DM). In a randomized clinical trial study, 46 T2DM patients, 30-70 years old recruited from "Diabetes Association of Iran-Babul ". Patients were randomly allocated to either the BJ group (n=23) who consumed 200 ml of BJ daily for eight weeks, or the control group (n=23) with no intervention. At the baseline and the end of 8-week intervention, blood pressure and biochemical markers were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose>100 mg/dL (5.6 mmol /L)
* Systolic blood pressure>130 mmHg or diastolic blood pressure>85mmHg
* Triglycerides> 150 mg/dL (1.7 mmol/L)

Exclusion Criteria:

* taking insulin
* smoking
* using antioxidant supplements

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-08-05 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose | 8 weeks
total cholesterol | 8 weeks

SECONDARY OUTCOMES:
LDL- cholesterol | 8 weeks
HDL- cholesterol | 8 weeks
Triglyceride | 8 weeks
HbA1c | 8 weeks
Systolic BP | 8 weeks
Diastolic BP | 8 weeks